CLINICAL TRIAL: NCT03680963
Title: Early Versus Differed Arterial Catheterization in Critically Ill Patients With Acute Circulatory Failure: A Multicentre, Open-label, Pragmatic, Randomised, Non-inferiority Controlled Trial (EVERDAC Trial)
Brief Title: Early Versus Differed Arterial Catheterization in Critically Ill Patients With Acute Circulatory Failure:
Acronym: EVERDAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR180137
Record Dates: First submitted 2018-09-11; First posted 2018-09-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Circulatory Failure
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive strategy (Experimental): Non-invasive strategy consisting of blood pressure monitoring by non-invasive automated cuff measurements
  Interventions: Procedure: Non-invasive strategy
- Control strategy (Other): Usual strategy of systematic indwelling arterial catheter insertion in the early hours of acute circulatory failure
  Interventions: Procedure: Control strategy

INTERVENTIONS:
Procedure: Non-invasive strategy — No indwelling arterial catheter insertion will be allowed during the first 28 days, excepted if predefined safety criteria (indicating absolute need of indwelling arterial catheter insertion) are reached.
  In the "non-invasive" group, automated oscillometric monitor will be used to monitor BP (blood pressure).
  Arms: Non-invasive strategy
Procedure: Control strategy — An indwelling arterial catheter will be inserted as soon as possible (within the first four hours after randomization) and will be maintained except in case of indwelling arterial catheter futility, suspected or proven indwelling arterial catheter related infection or thrombosis (at discretion of attending physician) until day 28 or ICU (Intensive Care Unit) discharge (whichever comes first). After day 28, clinicians may choose to maintain or to remove indwelling arterial catheter.
  Arms: Control strategy

SUMMARY:
The objective of the present research is a combination of a one-sided test of non-inferiority and a one-sided test of superiority. A stepped approach will be used to evaluate these hypotheses:

1. a less invasive intervention (i.e., no indwelling arterial catheter insertion until felt absolutely needed, according to consensual and predefined safety criteria) is non inferior to usual care (i.e., systematic indwelling arterial catheter insertion in the early hours of shock) in terms of mortality at day 28 (non-inferiority margin of 5%).
2. a less invasive intervention is not only non-inferior but also superior to usual care in terms of mortality.

Multi-centre, pragmatic, randomised, controlled, open, two-parallel group, non-inferiority clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years the day of inclusion
* Existence of an acute circulatory failure defined by the presence of the following items 1 and 2:

  1. Persisting hypotension (systolic blood pressure less than 90 mmHg or mean arterial blood pressure less than 65 mmHg) for more than 15 min at intensive care unit admission or within the following 24 hours, OR requirement of continuous intravenous vasopressor treatment (i.e. any dose of norepinephrine / epinephrine)
  2. Presence at least one of the following signs of hypoperfusion: alteration of mental status; skin mottling; oliguria defined as a urine output < 0.5 mL/kg body weight for at least one hour; arterial lactate > 2 mmol/L; peripheral venous lactate > 3.2 mmol/L; ScvO2 <70%
* Free express oral and informed consent of the patient or a proxy in case of impossibility for the patient to consent; emergency inclusion possible when legal representatives and patient's family are not available
* French health insurance holder

Exclusion Criteria:

* Acute circulatory failure, as defined by items 1 and 2 in inclusion criteria list (cf. supra) present for more than 24 hours
* Non invasive blood pressure (NIBP) device fails to display a blood pressure value, or cuff placement impossible
* Patient for whom an Extra-Corporeal Membrane Oxygenation (ECMO) therapy (either veno-arterial or venous-venous) is already in place or is to be initiated within the next 6 hours
* Patient treated with vasopressor doses of more than 2.5 μg/kg/min of norepinephrine tartrate plus epinephrine for at least 2 hours (i.e., for instance, more than 8 mg of norepinephrine tartrate in 50 mL at the rate of 66 mL/hour for a patient weighing 70 kg) (please note that in fact this dosage corresponds to 1.25 μg/kg/min of norepinephrine base)
* Severe traumatic brain injury (i.e., traumatic brain injury with a Glasgow coma scale score of less than 9 before sedation)
* Patient previously included in the trial
* Body mass index (BMI) above 40 kg/m2
* Pregnancy
* Brain death
* Moribund patient
* Patient known, at time of inclusion, as being under guardianship, authorship or curators

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
All-cause mortality by 28 days after randomisation | Patients will be followed from randomization to day 28

SECONDARY OUTCOMES:
To account for the potential bias brought by deaths occurring as the result of life-sustaining treatments withdrawal/withholding, as frequently encountered in intensive care unit, the investigators will record such events | From inclusion to Day 35
Cumulative incidence of death | From inclusion through Day 90
Cumulative survival free of indwelling arterial catheter insertion | From inclusion through Day 90
Number of patients who underwent indwelling arterial catheter insertion, in both groups | From randomization to Day 28
Evolution of daily Sequential Organ Failure Assessment (SOFA) score | During the first seven days
  The score (ranged from 0 to 24, the worth outcome) is based on six sub-scores (each ranged from 0 to 4, the worth outcome), one for each respiratory system, neurological, cardiovascular, hepatic, renal and coagulation.
Daily amount of intravenous fluid given for rapid vascular volume expansion | From Day 1 to Day 7
Duration of mechanical ventilation | From inclusion to Day 28
Ventilator-free days | From Day 1 to Day 28
  Patients dying between randomisation and Day 28 will be assigned a 0 value; for survivors at Day 28, all the days free of invasive mechanical ventilation through an endotracheal tube within the 28-day period will be taken into account
Proportion of patients treated by renal-replacement therapy | Between Day 1 and Day 28
Renal replacement therapy-free days | From Day 1 to Day 28
  Days without renal replacement therapy from Day 1 to Day 28 for survivors at Day 28, and from Day 1 to the date of death for patients dying before Day 28, will be taken into account
Proportion of patients treated by vasopressor | Between Day 1 and Day 28
Vasopressor therapy-free days | From Day 1 to Day 28
  Days without vasopressor therapy from Day 1 to Day 28 for survivors at Day 28, and from Day 1 to the date of death for patients dying before Day 28, will be taken into account
Mean daily blood volume drawn for lab testing during intensive care unit stay | From inclusion to Day 28
Number of blood cultures performed during intensive care unit stay | From inclusion to Day 28
Number of attempts at arterial puncture during intensive care unit stay | From inclusion to Day 28
Evolution of blood haemoglobin level | From Day 1 to Day 28
Evolution of haematocrit | From Day 1 to Day 28
Number of red blood cell packs transfused | From Day 1 to Day 28
Number of transcutaneous arterial and venous puncture for lab tests, arterial catheter insertion and set up of monitor, blood drawing from the arterial catheter or other vascular line | From inclusion to Day 28
Time (min) spent by nurses and physicians (min) on these tasks | During the first three days of the intensive care unit stay
  This outcome measure is planned to be collected during the first three days in a random sample of 10% of the study population and will be only considered during the medico-economic analyses.
Number of arterial and central venous catheter insertion during intensive care unit stay | From inclusion to Day 28
  Expressed as the incidence of new cases per 1000 catheter-days, including local and catheter-related bloodstream infections as consensually defined.
Numbers of arterial and central venous catheter-related infections | During intensive care unit stay
  Number of new cases per 1000 catheter-days
Numbers of local infections of arterial and central venous | During intensive care unit stay
  Number of new cases per 1000 catheter-days
Numbers of arterial and central venous catheter-related bloodstream infections | During intensive care unit stay
  Number of new cases per 1000 catheter-days
Number of bloodstream infections | During intensive care unit stay
Duration of intensive care unit stay | From inclusion to discharge
Duration of hospital stay | From inclusion to discharge
Intensive care unit mortality | From inclusion to discharge
Hospital mortality | From inclusion to discharge
Day 90 mortality | Day 90
Number of Adverse Events of special interest | From inclusion to Day 90
Incremental Cost-Effectiveness Ratio | At Day 28
Budget impact analysis of the generalization of the non-invasive strategy | on a 5 years' time frame
  The budget impact analysis will be to multiply the average annual cost per patient over 5 years by the number of eligible patients, taking into account a penetration rate
Pain related to the device used for blood pressure monitoring | Once a day, from inclusion to Day 28
  Numerical scale assessment of patient-reported pain related to the device used for blood pressure monitoring.
  Using the following 11-point numerical scales, ranged from 0 (no pain) to 10 (very important and permanent pain).
Discomfort related to device used for blood pressure monitoring | One a day, from inclusion to Day 28
  Numerical scale assessment of patient-reported discomfort related to the device used for blood pressure monitoring Using the following 11-point numerical scales, ranged from 0 (no discomfort) to 10 (very important and permanent discomfort).
Daily fluid balance of intakes and loss | The first seven days
  Difference between the daily amounts of:
  * daily fluid administration (in milliliter): intravenous hydration, vascular filling, enteral hydration
  * and the daily fluid loss (in milliliter): urine and fluid removal (during renal replacement therapy), tube drainage, estimated blood loss (laboratory test, bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire MULLER, Principal Investigator — UNIVERSITY HOSPITAL, ORLEANS
Locations (9):
- France (9):
  - Intensive care, Argenteuil
  - Intensive care, Dijon
  - Intensive care, La Roche-sur-Yon
  - Intensive care, Montauban
  - Intensive care, Nantes
  - Intensive care, Orléans
  - Intensive care, Poitiers
  - Intensive care, Strasbourg
  - Intensive care, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Muller G, Contou D, Ehrmann S, Martin M, Andreu P, Kamel T, Boissier F, Azais MA, Monnier A, Vimeux S, Chenal A, Nay MA, Salmon Gandonniere C, Lascarrou JB, Roudaut JB, Plantefeve G, Giraudeau B, Lakhal K, Tavernier E, Boulain T; CRICS-TRIGGERSEP F-CRIN Network and the EVERDAC Trial Group. Deferring Arterial Catheterization in Critically Ill Patients with Shock. N Engl J Med. 2025 Nov 13;393(19):1875-1888. doi: 10.1056/NEJMoa2502136. Epub 2025 Oct 29. PMID 41159885
- [Derived] Muller G, Kamel T, Contou D, Ehrmann S, Martin M, Quenot JP, Lacherade JC, Boissier F, Monnier A, Vimeux S, Brunet Houdard S, Tavernier E, Boulain T. Early versus differed arterial catheterisation in critically ill patients with acute circulatory failure: a multicentre, open-label, pragmatic, randomised, non-inferiority controlled trial: the EVERDAC protocol. BMJ Open. 2021 Sep 14;11(9):e044719. doi: 10.1136/bmjopen-2020-044719. PMID 34521655

DOCUMENTS (2):
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT03680963/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT03680963/SAP_001.pdf